CLINICAL TRIAL: NCT06397404
Title: Congestion Assessment Using Venous Excess Ultrasound Score (VExUS) in Patients With Acute Heart Failure
Brief Title: VExUS in Patients With Acute Heart Failure
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SS-DCFUD-02-2023
Record Dates: First submitted 2024-04-06; First posted 2024-05-02 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Heart Failure
Keywords: Cardiorenal Syndrome; Acute Kidney Injury; Fluid Overload; VEXUS; Natriuresis; Diuretics resistance; Congestion; Intrarenal blood flow
MeSH Terms: conditions — Cardio-Renal Syndrome; Acute Kidney Injury; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute decompensated heart failure: The study involved patients over 18 years of age admitted to the hospital with acute heart failure and requiring intravenous administration of loop diuretics. Diagnosis was based on the European Society of Cardiology (ESC) heart failure guidelines, with patients presenting with dyspnoea at rest or with minimal exertion and signs and symptoms of congestion (rales on chest auscultation, peripheral oedema, swelling of the cervical veins, hepatomegaly, ascites, hepatojugular reflux) and N-terminal pro-B-type natriuretic peptide (NT-proBNP) >1000 pg/ml.
  Interventions: Diagnostic Test: Venous excess ultrasound score (VExUS) protocol

INTERVENTIONS:
Diagnostic Test: Venous excess ultrasound score (VExUS) protocol — All patients upon admission undergo ultrasound assessment of diameter and collapsibility of the inferior vena cava, hepatic vein Doppler, portal vein Doppler, intra-renal venous Doppler.

SUMMARY:
The importance of assessing venous congestion in heart failure patients is widely acknowledged, but its study is hampered by the lack of a practical evaluation tool. Venous excess ultrasound score (VExUS) is a promising noninvasive ultrasound-guided modality that can detect and objectify clinically significant organ congestion. VExUS congestion grading score was still not formally validated in patients with AHF, as there is limited data on its clinical application in this group of patients.

DETAILED DESCRIPTION:
It is currently unknown whether changes in systemic venous congestion, assessed by venous excess ultrasound score (VExUS), are associated with worsening renal function, reduced diuretic and natriuretic response, and poor prognosis in patients with acute decompensation of heart failure (AHF).

This prospective, observational, single-center study included patients admitted to the intensive care unit with AHF. At admission all patients undergo bedside Doppler ultrasound of inferior vena cava, hepatic, portal and renal veins to determine blood flow patterns. Congestion was graded with the VExUS score (grade 0, grade 1, grade 2, grade 3). Sodium concentration in a spot urine sample was assessed in 1 hour after first standard intravenous loop diuretic administration. The primary endpoint was the development of acute kidney injury (AKI), defined as oligoanuria (diuresis rate <0.5 ml/kg/hour for 6 hours) and an increase of serum creatinine >26 µmol/l within a 48-hour period or 50% from baseline creatinine within a week. The secondary endpoints were in-hospital mortality, change in spot urine sodium content <50 mmol/l and development of diuretics resistance (defined as the need to double starting dose of intravenous furosemide in 6 hours without adding a different class of diuretic agents).

ELIGIBILITY:
Inclusion Criteria:

* Acute decompensation of heart failure (diagnosis was based on the European Society of Cardiology (ESC) heart failure guidelines, with patients presenting with dyspnoea at rest or with minimal exertion and signs and symptoms of congestion (rales on chest auscultation, peripheral oedema, swelling of the cervical veins, hepatomegaly, ascites, hepatojugular reflux) and N-terminal pro-B-type natriuretic peptide (NT-proBNP) > 1000 pg/ml

Exclusion Criteria:

* Chronic renal replacement therapy or glomerular filtration rate < 15 ml/min/1.73m 2 (chronic kidney disease Epidemiology Collaboration (CKD)-EPI)
* Cirrhosis with portal hypertension
* Acute myocardial infarction according to The Fourth Universal Definition of Myocardial infarction
* Pulmonary embolism
* Sepsis (according to The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3))
* Endotracheal intubation at the time of admission
* Pregnancy or breastfeeding
* Aortic dissection
* Active cancer
* Neurological or mental disease during exacerbation
* Refusal to sign an informed consent form, inadequate acoustic window

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involved patients over 18 years of age admitted to the hospital with AHF and requiring intravenous administration of loop diuretics. Diagnosis was based on the European Society of Cardiology (ESC) HF guidelines, with patients presenting with dyspnoea at rest or with minimal exertion and signs and symptoms of congestion (rales on chest auscultation, peripheral oedema, swelling of the cervical veins, hepatomegaly, ascites, hepatojugular reflux) and N-terminal pro-B-type natriuretic peptide (NT-proBNP) >1000 pg/ml.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Development of acute kidney injury (AKI) | During 7 days of hospital stay
  Assessment of patient's serum creatinine at admission, in 48 hours, at day 7, and calculation of the amount of urine output in the first 6 h after the administration of a loop diuretic.

SECONDARY OUTCOMES:
In-hospital mortality | During patient's hospital stay (up to 14 days)
  Death from any cause, whichever came first
Change in spot urine sodium content <50 mmol/l | 1 hour after first standard intravenous loop diuretic administration after patient's admission.
  Sodium concentration in a spot urine sample is assessed in 1 hour after first intravenous loop diuretic administration. Reduction of natriuretic response in the face of congestion with volume overload with spot urine sodium content <50 mEq/L generally identifies a patient with an insufficient diuretic response.
Development of diuretics resistance (defined as the need to double initial dose of intravenous furosemide in 6 hours without adding a different class of diuretic agents) | 6 hours after first intravenous furosemide administration
  Assessment of diuretic response: patient's urine output (ml/kg/hour) in the first 6 hours and patient's medical record with doses of administered diuretics.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Sovetova, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- City clinical hospital named after S. S. Yudin, Moscow City Health Department, Moscow, Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Local Ethics Committee policy

REFERENCES:
- See also: ACC Middle East & Eastern Mediterranean 2023, Athens, Greece, poster presentation. "Assessment of intrarenal venous flow can predict acute kidney injury in patients with acute heart failure." Sofia Sovetova — https://www.acc.org/-/media/Non-Clinical/Files-PDFs-Excel-MS-Word-etc/Meetings/2023/Agendas/ME-2023-Agenda.pdf
- See also: Sovetova, S, Andreev, D, Shchekochikhin, D. IMPACT OF RENAL BLOOD FLOW PATTERNS ON DIURETIC RESPONSE IN PATIENTS WITH ACUTE DECOMPENSATION OF HEART FAILURE. J Am Coll Cardiol. 2024 Apr, 83 (13_Supplement) 335 — https://doi.org/10.1016/S0735-1097(24)02325-8